CLINICAL TRIAL: NCT06243185
Title: A Phase II Study of the CDK4/6 Inhibitor Dalpiciclib Combined With Letrozole in Unresectable Refractory or Resistant Recurrent HR+/HER2 - Gynecologic Solid Tumors
Brief Title: Dalpiciclib Combined With Letrozole in HR+/HER2 - Gynecologic Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fengzhi Feng (Other)
Responsible Party: Sponsor-Investigator, Fengzhi Feng, professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K4823
Record Dates: First submitted 2024-01-09; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — dalpiciclib; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib+letrozole (Experimental): Drug: Dalpiciclib 150mg qd, d1-21, q4w Letrozole 2.5mg qd, q4w
  Interventions: Drug: Dalpiciclib plus letrozole

INTERVENTIONS:
Drug: Dalpiciclib plus letrozole — Dalpiciclib 150mg qd, d1-21, repeated once every 4 weeks. Letrozole 2.5mg qd, repeated once every 4 weeks.

SUMMARY:
This is a prospective, single-arm, single-center registry study to investigate 6-month progression-free survival with Dalpiciclib, a CDK4/6 kinase inhibitor, plus letrozole in patients with unresectable refractory or resistant recurrent HR-positive, HER2-negative gynecologic solid tumors." Dalpiciclib is a CDK4/6 kinase inhibitor that selectively inhibits the activity of CDK4/6 kinase, so that the complex with Cyclin D cannot phosphorylate the downstream Rb protein and prevent cells from entering the S phase from G1 phase, thereby inhibiting cell proliferation and anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years and ≤75 years;
2. Women with pathologically confirmed HR-positive, HER2-negative ovarian cancer or uterine tumors (including but not limited to high-grade serous ovarian cancer, low-grade serous ovarian cancer, ovarian endometrioid cancer, endometrioid cancer, low -grade endometrial stromal sarcoma, and uterine leiomyosarcoma) with evidence of focal recurrence or metastasis; Non-curative surgical resection or radiation therapy failing standard treatment, and no standard chemotherapy regimen. Er-positivity and/or PR-positive tumor cells were defined as 1% or more of all tumor cells that stained positively (as confirmed by the site investigator). Her2-negative was defined as 0/1+ on standard immunohistochemical (IHC) testing; An HER2/CEP17 ratio of less than 2.0 or a HER2 gene copy number of less than 4, as assessed by in situ hybridization (ISH), was confirmed by site investigator review.
3. Receipt of any previous systemic anticancer therapy for focal recurrent or metastatic disease.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Measurable lesions meeting RECIST 1.1 criteria or bone-only metastatic lesions (including osteolytic lesions or mixed osteolytic/osteogenic lesions).
6. Adequate organ and bone marrow function, defined as neutrophil count (ANC) ≥ 1500/mm3(1.5 × 109/L) (no growth factor administration within 14 days); Platelet count (PLT) ≥ 100,000/mm3 (100 × 109/L) (no corrective therapy within 7 days); Hemoglobin (Hb) ≥ 9 g/dL (90 g/L) (no corrective therapy used within 7 days); Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 60 ml/min; Total bilirubin (BIL) ≤ 1.5 times upper limit of normal value (ULN); Aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) ≤ 2.5 times The upper limit of normal (ULN), patients with liver metastases should be ≤ 5×ULN.
7. Use of a medically approved contraceptive method (e.g., an intrauterine device, contraceptive pill, or condom) during the study treatment period and for 3 months after the end of the study treatment period for patients with potential childbearing potential; A negative serum HCG test must have been performed within 72 hours before study entry; And had to be non-lactating.
8. All acute toxic effects prior to antineoplastic therapy resolved to grade 0-1 (according to NCICTCAE version 5.0) or to the level specified in the inclusion/exclusion criteria. Other toxicities, such as alopecia, that were deemed by the investigators not to pose a safety risk to patients were excluded.
9. There is no limit to the number of previous lines of endocrine therapy.
10. The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Previous pathological diagnosis of HER2-positive. Patients who were not candidates for endocrine therapy as judged by the investigator. "Patients were included who were symptomatic, had spread to the viscera, and were at risk for life-threatening complications in the short term (including patients with uncontrolled massive exudates [thoracic, pericardial, abdominal], pulmonary lymphangitis, and more than 50% liver involvement)." 3.Patients with brain metastases diagnosed by head CT or MRI. 4.Patients had received any previous CDK4/6 inhibitor therapy. 5.Major surgery, chemotherapy, radiation therapy, any investigational drug, or other anticancer treatment within 2 weeks before study entry.

6.Any other malignancy was diagnosed within 3 years before study entry, except nonmelanoma skin cancer, basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix treated with curative intent 7.Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥1000 IU/ml), hepatitis C (positive hepatitis C antibody and HCV-RNA higher than the lower limit of detection of the assay), or co-infection with hepatitis B and C.

8.In the 6 months prior to study entry, the following occurred: Myocardial infarction, severe

or unstable angina, cardiac dysfunction of NYHA class 2 or higher, persistent arrhythmia of class 2 or higher (according to NCICTCAE, version 5.0), atrial fibrillation of any grade, coronary or peripheral artery bypass grafting, symptomatic congestive heart failure, or cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism).

9.Severe infection (e.g., intravenous antibiotics, antifungal, or antiviral agents according to standard practice) within 4 weeks before the first dose or unexplained fever >38.5oC during screening/before the first dose.

10.Inability to swallow, intestinal obstruction, or other factors affecting drug administration and absorption.

11.Known allergies to letrozole or anastrozole, LHRH agonist (goserelin), SHR6390/ placebo, or any excipients.

12.Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

13.Known history of psychotropic drug abuse or drug use. 14.Patients with other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study or interfere with the study results, and those who are considered by the investigator to be unsuitable for participation in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | From the start of randomization to 6 months
  according to RECIST1.1 criteria,the percent of participant whose PFS is more than 6 months

SECONDARY OUTCOMES:
Progression-free survival(PFS) | From the start of randomization to a minimum of 1 year
  Time from initiation of study protocol treatment to disease progression or death
Objective Response Rate（ORR） | From the start of randomization to a minimum of 1 year
  Percentage of patients with CR/PR in the number of patients that whose tumour can be evaluated.
Disease Control Rate (DCR) | From the start of randomization to a minimum of 1 year
  Percentage of patients with CR/PR/SD in the number of patients that whose tumour can be evaluated.
Duration of response（DOR） | From the start of randomization to a minimum of 1 year
  The time between the onset of efficacy and confirmation of tumor progression
Overall Survival(OS) | up to 2 years
  The time from the start of treatment with this study protocol to the time of all-cause death of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi f Feng, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided